CLINICAL TRIAL: NCT04575324
Title: Project STAMINA (Syringe Service Telemedicine Access for Medication-assisted Intervention Through NAvigation): Development and Testing of a Health Navigation Approach for Linking Syringe Service Program Clients to Medication Assisted Treatment
Brief Title: Project STAMINA (Syringe Service Telemedicine Access for Medication-assisted Intervention Through NAvigation)
Acronym: STAMINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1138-0420
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Opioid-use Disorder
Keywords: Opioid Use Disorder; Injection Drug Use; Telemedicine; Telehealth; Syringe Exchange; Medication for Opioid Use Disorder; Medication Assisted Treatment; Substance Use Disorder; Syringe Service Program; Needle Exchange
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will receive the telemedicine linkage intervention.
  Interventions: Behavioral: Telemedicine Linkage Intervention
- Control Arm (No Intervention): Participants will receive a standard referral to an in-person MOUD treatment appointment, which typically occurs within 24-72 hours. They also receive a bus pass to cover transportation (both directions), as well as an appointment reminder card.

INTERVENTIONS:
Behavioral: Telemedicine Linkage Intervention — Participants will be immediately linked to telemedicine care provided by an FQHC provider waivered to prescribe buprenorphine and naltrexone or able to refer patients to methadone treatment. Participants will have their vitals checked and be virtually connected to the provider. The research assistant will share the vitals with the provider, and the provider will provide personalized care during which they discuss treatment options with the participant. If a medication for opioid use disorder is prescribed or if a methadone referral is made, transportation assistance will be provided to the participant as part of the intervention. Transportation to pick up the prescription or complete the first appointment will be provided via a HIPAA compliant ride-share company, and a bus pass will be provided to the participant for the return trip.
  Arms: Intervention Arm

SUMMARY:
Project STAMINA is a clinical trial that seeks to establish effectiveness of a telemedicine approach for linking syringe exchange clients to medications for opioid use disorder. This pilot study aims to recruit n=275 people and utilizes two study arms: (1) a treatment arm consisting of immediate telemedicine linkage and (2) a control arm consisting of standard referral to treatment. Half of the study participants will be randomly enrolled in each arm. The study will utilize qualitative and quantitative data, including questionnaire data, drug test results, and administrative treatment data, at multiple time points to determine what effect telemedicine linkage has on clients in relation to the comparison group.

DETAILED DESCRIPTION:
INTERVENTION DESCRIPTION:

Project STAMINA utilizes two study arms: (1) a treatment arm consisting of immediate telemedicine linkage (2) a control arm consisting of standard referral to treatment. Half of the study participants will be randomly enrolled in each arm. All enrollment and telemedicine care will occur at one of two Chicago-based and university-affiliated syringe service program (SSP) sites, where the primary purpose is providing free access to syringes for people who inject drugs.

Intervention Arm (1): Participants enrolled into the telemedicine linkage intervention will be immediately linked to telemedicine care provided by a university-affiliated federally qualified health center (FQHC) that can prescribe buprenorphine and naltrexone and has a relationship with a methadone treatment provider they can refer patients to as appropriate. Study participants prescribed buprenorphine or naltrexone will be able to receive MOUD treatment at any of the 6 FQHC locations across the city, three of which are in relatively close proximity to the SSP sites, and a no-cost induction buprenorphine prescription can be dispensed from their main office. The FQHC can also refer to a methadone provider with various locations throughout the city. At the SSP, the participant will have their vitals checked by a research team member and be connected with the FQHC provider via an iPad. The research assistant will share the participant's vitals with the provider, and the provider will complete a virtual treatment appointment. The research assistant will offer the participant transportation assistance to pick up the first buprenorphine or naltrexone prescriptions or to attend the first methadone referral appointment. Transportation to pick up the prescription will be provided via a HIPAA compliant ride-share company, and a bus pass will be provided to the participant for the return trip. Further, to support the intervention, the research assistant will also provide a visual guide at enrollment (i.e. picture directions) that describes how to navigate the FQHC pharmacy, as well as a scheduling card that allows them to record any MOUD appointment dates. All follow-up OUD care and prescribing will be conducted based on the provider's standards and may include in-person or telemedicine appointments.

Standard Care Arm (2): Participants enrolled in the control arm will receive a standard referral to an in-person appointment, also with a provider from the same FQHC sites or a methadone provider of their choice. This appointment will involve an in-person meeting with the provider, which will occur within 24-72 hours of the enrollment time. After study enrollment, the research assistant will schedule this in-person appointment. The research assistant will also provide the participant with an appointment reminder card for this appointment and bus passes to cover the transportation to and from the appointment, which aligns with standard care at the SSP. All follow-up OUD care and prescribing will be conducted based on the provider's standards and may include in-person or telemedicine appointments.

RESEARCH DESIGN:

Participants will be identified one of the following ways: (1) individuals will see the STAMINA poster within the syringe exchange sites and be able to ask staff where to get more information, (2) current syringe service clients will be able to inform staff that they are interested in treatment for an opioid use disorder, and staff will inform them of the study opportunity, (3) individuals will be able to see STAMINA flyers at other social service programs in the city or on social media platforms and be able to call study personnel for more information on study enrollment, or (4) individuals will be introduced to the study by street outreach staff.

Research personnel will be responsible for assessing individuals for eligibility. Using the recruitment script, after providing an introduction to STAMINA and a reason for the eligibility questions, the research assistant will begin to read the full script, which includes an assessment of eligibility criteria. Any client who is eligible and interested in participating will move forward with the statement of informed consent. Willing participants will be asked to sign the consent form. Once the participant has been officially enrolled, the onsite research assistant will notify an offsite research assistant of the enrollment so that the participant can be randomized. This allows the onsite research assistant to move forward in collecting data while blinded to the study arm assignment.

This offsite research assistant will use the pre-established random arm assignment list to determine which arm the client has been randomly assigned, based on their study identification number. Each identification number will include two stratified randomization blocks: (1) one arm assignment will be for participants who are interested in receiving buprenorphine or naltrexone, or open to considering these types, [Open MOUD Stratified Arm Assignment] (2) one arm assignment will be for participants who are only interested in receiving methadone [Methadone Only Stratified Arm Assignment]. Based on the participant's interest in MOUD, which will have been clarified during the eligibility assessment and entered into the data collection system, the offsite research assistant will then read the appropriate random arm assignment from the list and record their random arm assignment in the data collection system. If the participant is assigned to the telemedicine intervention arm, the offsite research assistant will need to notify the FQHC of an upcoming virtual appointment [the FQHC needs a one-hour notice of appointment]. At this time, the offsite research assistant will not yet inform the onsite research assistant, or the participant, of the arm assignment so that baseline data collection can be completed prior to notification.

The onsite research assistant will be responsible for data collection. The first step in data collection will be to complete a questionnaire. The questionnaire will take approximately 45-60 minutes and be administered by research staff using the Research Electronic Data Capture (REDCap) data collection system, which is a secure, HIPAA-compliant, web-based survey instrument. The questionnaire will be administered in a standard manner, meaning: (1) all questions will be asked, (2) all questions will be read as written, (3) research assistants will not reword questions in any way, and (4) participants have the right to refuse to answer any question.

This questionnaire will cover the following topics:

* Full name, Date of Birth, SSN, and UI Health Medical Record Number (MRN)
* Demographic information
* Social support
* Child welfare involvement
* Housing and homelessness
* Alcohol use
* Drug use
* Heroin cravings
* Opioid withdrawal symptoms
* Overdose experiences
* Physical and mental health
* Trauma exposure
* Criminal justice involvement
* Treatment motivation
* Quality of life

The questionnaire will also request participant contact information. This information will not be used as research data, but rather, will aid the scheduling of research follow-up visits. The form will ask participants for (1) their contact information, (2) the contact information for others who might be able to help in reaching the participant, (3) the contact information for providers whose services they utilize and might be able to help reach the participant. The participants are reminded at the beginning of the form that they have the right to refuse any question and only share what they want to share. Because of the transient nature of the participant population, additional contacts are helpful in reaching the participant should personal contact information change.

Participants will be asked to complete the REDCap questionnaire at baseline and 3 months after baseline. Each questionnaire will take 45-60 minutes to complete. Depending on participant availability, the follow-up questionnaire (3-months) will be completed by a research team member at the SSP site or by telephone.

In addition to the questionnaire, all participants will be asked to submit a urine drug screen at baseline and 3-months as a form of data collection. The drug screen will be completed on-site at the SSP and takes 1-2 minutes to complete. When possible, even if a participant completes the questionnaire by telephone, they will still be asked to return to the SSP within 24 hours of completing their questionnaire to complete the follow-up drug screen.

At baseline, once participants have completed all data collection, they will be notified of their random study arm assignment. At this time, participants randomized to the telemedicine intervention arm would be connected via telemedicine to the FQHC provider and take part in the intervention described above. Participants randomized to the control arm would receive a scheduled in-person appointment.

At the end of the visit with the research staff, all participants will receive materials that aid follow-up data collection and prepare them for the data collection timeline. All participants will be given a scheduling form that visually displays the data collection items in the order of their occurrence. Participants will also be provided with the STAMINA contact telephone number and asked to store it in their phone, if applicable.

SECONDARY DATA COLLECTION:

As a part of the consent and health information release process, we request to access participant protected health information (PHI) from the four sources listed below.

(1) FQHC and (2) methadone provider We will request that the FQHC and methadone provider pull treatment data, including dates of service, medications prescribed, and treatment details to understand compliance.

(3) State Prescription Monitoring Program (PMP) records We will request the state prescription monitoring program (PMP) data for the purpose of verifying the information provided by the participant during the REDCap questionnaire. While we ask the participant to self-report whether they have engaged in medication for opioid use disorder treatment, the PMP data will allow us to verify whether they have been prescribed/dispensed any of the prescriptions or prescriptions not mentioned during the interview.

(4) State Vital Records Similarly, we request state vital records data for the purpose of verifying whether a participant passed away. We are obtaining this data to verify if a participant disengaged from the study because of death and to understand whether that death was caused by drug use.

ELIGIBILITY:
Inclusion Criteria:

* communicate in English
* be at least 18 years of age
* reside in Cook County, Illinois
* score at least "2" on the Opioid Use Disorder Screening tool (DSM), indicating mild opioid use disorder
* express interest in receiving medication for an opioid use disorder (MOUD)

Exclusion Criteria:

* have plans to move outside of Cook County, Illinois within the next 6 months
* have plans to serve a sentence that requires reporting to jail or prison within the next 6 months
* score "36" or higher on the Clinical Opioid Withdrawal Scale (COWS), indicating severe opioid withdrawal symptoms
* currently taking any form of medication that has been prescribed by a healthcare provider to treat opioid use disorder
* demonstrate inadequate ability to provide informed consent, as indicated by poor understanding of research based on 3 competency questions asked related to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Watson, PhD, Principal Investigator — Chestnut Health Systems; James A Swartz, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Community Outreach Intervention Projects (COIP) Field Site, Chicago, Illinois, United States

REFERENCES:
- [Derived] Franceschini D, Swartz JA, Watson DP, Mackesy-Amiti ME, Taylor L, Zhao P, Messmer S, Jimenez AD, Gastala N. Syringe Service Program-Based Telemedicine Linkage to Opioid Use Disorder Treatment: Results From a Pragmatic Randomized Trial of the STAMINA Intervention. Subst Use. 2025 Nov 24;19:29768357251372336. doi: 10.1177/29768357251372336. eCollection 2025 Jan-Dec. PMID 41306931
- [Derived] Watson DP, Ray B, Phalen P, Duhart Clarke SE, Taylor L, Swartz J, Gastala N. Fentanyl Exposure and Detection Strategies Utilized by Clinical Trial Participants Seeking Linkage to Opioid Use Disorder Treatment at a Syringe Service Program. J Med Toxicol. 2024 Jan;20(1):13-21. doi: 10.1007/s13181-023-00979-7. Epub 2023 Dec 4. PMID 38048033
- [Derived] Watson DP, Swartz JA, Robison-Taylor L, Mackesy-Amiti ME, Erwin K, Gastala N, Jimenez AD, Staton MD, Messmer S. Syringe service program-based telemedicine linkage to opioid use disorder treatment: protocol for the STAMINA randomized control trial. BMC Public Health. 2021 Mar 31;21(1):630. doi: 10.1186/s12889-021-10669-0. PMID 33789642

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 138 (Enrolled and completed baseline interview) | 137 (Enrolled and completed baseline interview)
Completed | 108 (Completed 3-month follow-up interview) | 109 (Completed 3-month follow-up interview)
Not Completed | 30 | 28
Not completed — Lost to Follow-up | 29 | 25
Not completed — Death | 1 | 2
Not completed — Withdrawn: Did not meet eligibility criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is N=274. This includes all 138/138 enrolled in the intervention arm and 136/137 enrolled in the control arm. One control arm participant was removed from the baseline analysis population as they were withdrawn from the study for not meeting eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.59 (10.15) | 48.92 (10.58) | 48.24 (10.37)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 106 | 107 | 213
  Female | 32 | 28 | 60
  Transgender | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 109 | 105 | 214
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 83 | 82 | 165
  White | 47 | 44 | 91
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 138 | 136 | 274
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 107 | 97 | 204
  Other | 31 | 39 | 70
Housing Status [Count of Participants; unit: Participants]
  Stable | 76 | 75 | 151
  Unstable | 62 | 61 | 123
Insurance Status [Count of Participants; unit: Participants]
  Uninsured | 18 | 18 | 36
  Insured | 115 | 113 | 228
  Unknown | 5 | 5 | 10
Syringe Exchange Client Status [Count of Participants; unit: Participants] — Whether clients had previously used the services of the syringe service sites.
  Participants
    No | 92 | 90 | 182
    Yes | 46 | 46 | 92
Prior Lifetime Overdose(s) [Mean (Standard Deviation); unit: overdoses] | 4.85 (10.86) | 3.80 (9.21) | 4.33 (10.07)
Opioid Use Severity [Mean (Standard Deviation); unit: units on a scale] — Opioid use severity was measured using the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Clinical Diagnostic Criteria for Opioid Use Disorder.
  Participants provided yes (1)/ no (0) responses to a series of 11 questions regarding the presence of symptoms associated with opioid use disorder in the past 12 months.
  The minimum value is 0, and the maximum value is 11. The severity of the opioid use disorder is defined as Mild (2-3 symptoms present), Moderate (4-5 symptoms present), or Severe (6 or more symptoms present).
  units on a scale | 10.48 (1.19) | 10.40 (1.05) | 10.44 (1.12)
Withdrawal Severity [Mean (Standard Deviation); unit: units on a scale] — Opiate withdrawal severity was measured using the Clinical Opiate Withdrawal Scale (COWS).
  Staff used observation to rate participants from (0-4) or (0-5) on 11 items representing commons symptoms of opiate withdrawal. The instrument is designed to utilize clinician observation; however, modifications were made to items # 2,5-7,10 to also question whether participants experienced the listed symptom (yes/no).
  The minimum value is 0, and the maximum value is 48. The severity of withdrawal is defined as Mild (5-12), Moderate (13-24), Moderately Severe (25-36), or Severe (more than 36).
  units on a scale | 5.00 (5.16) | 4.00 (3.74) | 4.50 (4.53)
Block Randomization [Count of Participants; unit: Participants] — Participants were asked during enrollment, prior to randomization, whether they are (1) willing to discuss all medication options with a provider ("MOUD open") or (2) only interested in methadone treatment ("Methadone only"). Population: Block randomization was added to the study protocol after 3 participants had been previously enrolled; thus, only 271 participants are included in this analysis population.
  Participants
    number analyzed (Participants) | 136 | 135 | 271
    MOUD open | 64 | 60 | 124
    Methadone only | 72 | 75 | 147

OUTCOME MEASURES:

1. Primary Outcome: Linkage to Medication for Opioid Use Disorder (MOUD)
Description: Whether the participant attends 1 in-person MOUD treatment appointment
Time Frame: Within 14 days of enrollment
Population: The analysis population is N=274. This includes all 138/138 enrolled in the intervention arm and 136/137 enrolled in the control arm; one control arm participant was removed from the outcome analysis population as they were withdrawn from the study for not meeting eligibility criteria. Electronic health record data were obtained for all 274 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 138 | 136
Participants
  Yes | 25 | 47
  No | 113 | 89

2. Secondary Outcome: Medication for Opioid Use Disorder (MOUD) Treatment Engagement
Description: Whether the participant attends 2 in-person treatment appointments
Time Frame: Within 34 days of enrollment
Population: The analysis population is N=274. This includes all 138/138 enrolled in the intervention arm and 136/137 enrolled in the control arm; one control arm participant was removed from the outcome analysis population as they were withdrawn from the study for not meeting eligibility criteria. Electronic health record data and prescription drug monitoring program data were obtained for all 274 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 138 | 136
Participants
  Yes | 19 | 29
  No | 119 | 107

3. Secondary Outcome: Medication for Opioid Use Disorder (MOUD) Treatment Retention
Description: Whether the participant is actively engaged in treatment (i.e. participant goes no more than 14 days without medication for opioid use disorder (MOUD) or being discharged from care)
Time Frame: 3 month study period
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 138 | 136
Participants
  Yes | 12 | 14
  No | 126 | 122

4. Secondary Outcome: Self-report Non-medication for Opioid Use Disorder (MOUD) Opioid Use
Description: Self reported days of non-prescribed opioid use in the past 30 days using questions from the National Survey on Drug Use and Health, which was modified to ask about separate known use of heroin, fentanyl/carfentanyl, and prescription pain killers
Time Frame: 3 month study period
Population: The analysis population is N=219. This includes only participants that completed a 3-month follow-up interview.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 110 | 109
Days | 19.09 (12.72) | 19.92 (12.08)

5. Secondary Outcome: Detected Non-prescribed Opioids
Description: Whether illicit opioids were detected through urine tests administered at 3 months.
Time Frame: 3 month study period
Population: The analysis population is N=149. This includes only participants that submitted a urine drug screen at the 3-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 73 | 76
Participants
  Yes | 52 | 56
  No | 21 | 20

ADVERSE EVENTS:
Time Frame: All-cause mortality data were collected for a duration of 6 months post-enrollment via the County's Medical Examiner records. All other adverse event and serious adverse event data were collected 3 months post-enrollment via follow-up interviews with participants.
Description: The total number of participants at risk for all-cause mortality is N=274. This includes 138/138 enrolled in the intervention arm and 136/137 enrolled in the control arm; one control participant was withdrawn for not meeting eligibility criteria and removed from monitoring. Medical Examiner records were searched for all 274 participants.
  The total number of participants at risk for all other adverse events is N=217. This includes only participants that completed a 3-month follow-up interview.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 2/138 | 2/136
Serious Adverse Events (participants affected / at risk) | 34/108 | 22/109
Other Adverse Events (participants affected / at risk) | 50/108 | 41/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=108) | Control Arm (N=109)
Drug Overdose (Injury, poisoning and procedural complications) | 19 | 19 — Reported at least 1 drug overdose
Suicide Attempt (Psychiatric disorders) | 7 | 2 — Reported at least 1 suicide attempt
Drug Overdose-Related Emergency Room Visit (Injury, poisoning and procedural complications) | 14 | 14 — Reported at least 1 drug overdose-related emergency room visit
Drug Overdose-Related Hospitalization (Injury, poisoning and procedural complications) | 3 | 3 — Reported at least 1 drug overdose-related hospitalization
Mental Health-Related Hospitalization (Psychiatric disorders) | 12 | 4 — Reported at least 1 mental health-related hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=108) | Control Arm (N=109)
New Chronic Health Condition (General disorders) | 33 | 29 — Reported at least 1 new chronic health condition
Mental Health-Related Outpatient Treatment (Psychiatric disorders) | 14 | 9 — Reported at least 1 mental health-related outpatient treatment
Criminal Arrests, Bookings, Charges (Social circumstances) | 12 | 7 — Reported at least 1 criminal arrest, booking, or charge
Criminal Detainment or Imprisonment (Social circumstances) | 12 | 4 — Reported at least 1 criminal detainment or imprisonment

LIMITATIONS AND CAVEATS:
The internal validity of the results of the study are restricted by the study's use of a pragmatic approach and limited control over the intervention and clients' MOUD treatment. Though our goal was to ensure generalizability and sustainability of the intervention, providing participants with autonomy over their methadone provider resulted in missing administrative data as data use agreements were only established with our FQHC partner and the city's largest methadone provider.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT04575324/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04575324/ICF_001.pdf